CLINICAL TRIAL: NCT05634265
Title: Social Media for ART Adherence and Retention in Adolescents and Young Adults: the Vijana-SMART Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Keshet Ronen, Assistant Professor, Global Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002554
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: HIV-1-infection; Adherence, Medication; Depression
MeSH Terms: conditions — Medication Adherence; Depression

STUDY DESIGN:
Intervention Model Description: Single-group pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot (Experimental): Participants will be offered the Vijana-SMART WhatsApp group intervention
  Interventions: Behavioral: Vijana-SMART

INTERVENTIONS:
Behavioral: Vijana-SMART — The Vijana-SMART intervention is a facilitated peer group, delivered through WhatsApp. Intervention messages were developed based on findings from formative interviews and social support theory, which posits that individuals experience social support through informational, instrumental, companionship and emotional forms. Groups will have approximately 25 members and will be facilitated by a study team member, by sending weekly scheduled messages, answering participant questions, and encouraging group discussion. Intervention messages were designed based on guidance from formative interviews; topics include ART adherence, medication side effects, nutritional practices, depression, social support, HIV status disclosure, stigma, positive prevention, substance use, and contraception.

SUMMARY:
The goal of this study is to investigate whether a virtual peer support group improves ART knowledge, adherence, and mental health in youth living with HIV in Kenya.

DETAILED DESCRIPTION:
Adolescents and young adults (AYA) living with HIV show lower ART adherence, higher loss to follow-up and higher AIDS-related mortality than other age groups. Innovative approaches are needed that address AYA's unique needs and improve their adherence and retention in HIV care. There is evidence that peer support and mobile messaging with healthcare workers (HCW) are two strategies that may be effective in this group, but their evaluation has been limited and no interventions have combined them. Since 2014, youth-run virtual support groups have spontaneously started at HIV clinics, using the mobile social media application WhatsApp. These groups present valuable case studies from which the proposed project will develop a structured social media intervention that combines peer and HCW support to improve ART adherence and retention, guided by the preferences of AYA. The SPECIFIC AIMS are to (1) Characterize the existing WhatsApp groups through in-depth interviews with members and detailed content analysis of the group's communications during a 6-week observation period. This will define the elements and features desired by AYA in a social media intervention. (2) Guided by findings from Aim 1, behavioral theory, and the study team's ongoing research on mobile messaging to improve ART adherence, to develop and refine structured content for a reproducible WhatsApp intervention that incorporates peer and HCW interaction. (3) Pilot the structured intervention for 6 months in another clinic and evaluate its impact on intermediate outcomes ART knowledge, depression and stigma.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* On ART
* Aware of HIV status
* Has access to WhatsApp
* Literate

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
ART information, motivation, behavioral skills | 6 months
  Self-reported score on abbreviated Lifewindows IMB instrument
Social support | 6 months
  Self-reported score on SS-B instrument
Stigma | 6 months
  Self-reported score on abbreviated ALHIV-SS instrument
ART adherence | 6 months
  Self-reported score on Wilson 3-item scale
Depression symptoms | 6 months
  Self-reported score on PHQ-9 scale
Resilience | 6 months
  Self-reported score on abbreviated Connor-Davidson scale

CONTACTS AND LOCATIONS:
Overall Officials: Keshet Ronen, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Kayole, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be posted to the Harvard Dataverse
Time Frame: Upon publication of results
Access Criteria: Data may not be used for profit

REFERENCES:
- [Derived] Ronen K, Mugo C, Kaggiah A, Seeh D, Kumar M, Guthrie BL, Moreno MA, John-Stewart G, Inwani I. Facilitated WhatsApp Support Groups for Youth Living With HIV in Nairobi, Kenya: Single-Arm Pilot Intervention Study. JMIR Form Res. 2023 Nov 13;7:e49174. doi: 10.2196/49174. PMID 37955957